CLINICAL TRIAL: NCT05206305
Title: Sensory-Evoked Cortical Gamma Oscillation: Impact on Visual Processing and Cognitive Function in Patients With Alzheimer's Disease
Brief Title: Sensory-Evoked Cortical Gamma Oscillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALD-001-122021
Record Dates: First submitted 2021-12-17; First posted 2022-01-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD Patients (Experimental): Patients with Alzheimer's Disease, as verified by positive A(beta)-PET and/or CSF tau/A(beta) biomarkers, who will receive one hour daily gamma frequency sensory stimulation from the investigational device for an 8 week period.
  Interventions: Device: GammaSense Stimulation device

INTERVENTIONS:
Device: GammaSense Stimulation device — Cognito Therapeutics GammaSense Stimulation device delivers sensory (auditory and visual) stimuli at a rate of 40 Hz to the wearer for one hour each day.

SUMMARY:
The purpose of the study is to investigate the efficacy of cortical gamma oscillation on visual sensory processing and cognitive function in Alzheimer's Disease (AD) patients by combining a therapeutic sensory stimulation device capable of evoking 40-Hz gamma oscillation via non-invasive visual and auditory stimulation with pre-established markers of cortical network activity, i.e., electroencephalography (EEG) and event-related potentials (ERP), to evaluate the applicability of the 40-Hz multimodel sensory stimulation as a novel therapeutic approach for treatment of AD patients.

DETAILED DESCRIPTION:
The central hypothesis of the study is that sustained 40Hz gamma oscillatory sensory stimulation therapy will improve cognitive function in patients with AD. The further hypothesis is that the improvement in cognitive function will result from improved connectivity and cortical network function as measured by EEG and ERP.

The hypotheses will be tested by the following:

1. - Elucidate the immediate impact of gamma oscillations on sensory processing and cognitive function by assessing cognitive function and cortical network function prior to the introduction of sensory stimulation and comparing it to post-therapeutic assessments immediately following the acute administration of therapy on visual processing.
2. - Explore the short and long-term therapeutic benefits of a sub-chronic (8 weeks) treatment by assessing cognitive function and cortical network connectivity immediately after the 8 week sensory stimulation therapy. If significant changes are observed between pre-therapy and post-therapy neurophysiologic data for an individual subject, neurophysiological testing will be repeated 4 weeks following the conclusion of therapy.
3. - Investigate the correlation between neurophysiology and cognitive function by assessing cognitive function and neurophysiological measures of cortical network activity at multiple time points to determine if therapeutic changes in one domain reflect changes related to the other domain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 60 and older with established diagnosis of Alzheimer's Disease as defined by the current consensus criteria for AD (Albert et al, 2011, Jack et al, 2011; McKhann et al, 2011)
* Fluent and literate in English language
* Able to consent for themselves based upon the MacArthur Competence Assessment Tool for Clinical Research
* Patients with a pre-existing positive A(beta)-PET and/or CSF tau/A(beta) markers or willingness to undergo a Lumbar Puncture (LP) with these results

Exclusion Criteria:

* Not fluent and literate in English
* Severe dementia
* Other medical conditions/neurodegenerative disease that could significantly impair cognitive abilities
* Cardiac pacemakers or any other implants that may not be compatible with MRI
* Cognitively impaired to the point the patient is unable to consent for themselves
* Claustrophobic to the point that medication is required

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cortical Network Functioning | 8 weeks
  Cortical visual processing assessed before and after first therapy session to evaluate immediate impact of therapy device on cortical network functioning. The same measurements will be applied again at the conclusion of 8 week therapy period to evaluate impact of the therapy device on cortical network functioning over the total study period.
Cognitive Status | 8 weeks
  Neuropsychological tests administered before & after 8 week therapy period. Aggregate scoring: Range 1-4. 1=All scores better than normal. 2=All scores normal. 3=1-2 scores abnormal 4=3+ scores abnormal. Tests administered are:
  * Montreal Cognitive Assessment (MoCA) tests memory, attention, language. Score range 0-30.
  * Craft Story 21 Recall (Immediate and Delayed) tests memory. Score range 0-44.
  * Benson Complex Figure (Copy and Recall) tests memory, visuospatial perceptive, fine-motor coordination. Score range 0-17.
  * Number Span (Forward and Backward) tests memory. Score range 0-14.
  * Category Fluency (Animals and Vegetables) tests verbal fluency, semantic memory. Score range 0-77.
  * Trail Making (A and B) tests visuomotor and perceptual scanning abilities. Score range 0-150 A (numerical sequence) & 0-300 B (letter sequence).
  * Multilingual Naming test (MINT) tests naming impairment. Score range 0-32.

SECONDARY OUTCOMES:
Resting state functional magnetic resonance imaging | 8 weeks
  Resting state fMRI performed before and after the 8 week therapy. Imaging will be compared to evaluate the impact of the investigational device on resting state cerebral network function

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fernandez-Romero, MD, Principal Investigator — University of Tennessee Medical Center
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No